CLINICAL TRIAL: NCT06421012
Title: Preoxygenation for Tracheal Aspirations in Intensive Care, a Randomized Controlled Trial
Brief Title: Preoxygenation for Tracheal Aspirations in Intensive Care
Acronym: POXTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230486; 2023-A00694-41 (Other: ANSM)
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: ICU Patients Under Invasive Mechanical Ventilation
Keywords: Endotracheal suctioning; Preoxygenation; Ventilation; ICU
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without additional preoxygenation (Experimental)
  Interventions: Procedure: Experimental : Patients without additional preoxygenation
- Patients with additional preoxygenation (Active Comparator)
  Interventions: Procedure: Active Comparator : Patients with additional preoxygenation

INTERVENTIONS:
Procedure: Experimental : Patients without additional preoxygenation — Throughout the entire period of their mechanical ventilation, patients will not receive additional preoxygenation before any endotracheal suctioning; their FiO2 value will be maintained constant
  Arms: Patients without additional preoxygenation
Procedure: Active Comparator : Patients with additional preoxygenation — Throughout the entire period of their mechanical ventilation, patients will receive additional preoxygenation at 100% FiO2 for a systematic 2-minute duration prior to any endotracheal suction. Subsequently, the FiO2 will be reset to the previous default value.
  Arms: Patients with additional preoxygenation

SUMMARY:
Clearing the airways is a complex phenomenon involving the production of secretions, the nature of mucus (viscosity, elasticity, stringiness, and adhesiveness), ciliary movement, and coughing. In intubated and ventilated patients, endotracheal suctioning occur when the patient is "unable to clear the airways of obstructions hindering the free passage of air." These suctioning can lead to transient desaturation exacerbated by a decrease in cardiac output due to increased mean arterial pressure, promoting cardiac arrhythmias. To minimize these effects, it is recommended to perform additional preoxygenation, by increasing the fraction of O2 in the air delivered to the patient by the ventilator 2-3 minutes before the procedure. These longstanding recommendations were reiterated in 2022, based on outdated studies involving systematic suctioning that required disconnecting the patient from the ventilator.

Currently, suctioning are performed on-demand, based on the patient's congestion status, either through the endotracheal tube cap or a "closed system." Desaturations have become infrequent without establishing that additional preoxygenation can prevent them. Moreover, additional preoxygenation is not without risks. By inducing de-nitrogenation atelectasis with a loss of lung volume, it can exacerbate pre-existing lung injuries in the most severe patients. In less severe cases, preoxygenation leads to transient hyperoxia, with various deleterious effects impacting patient prognosis. Thus, a short-term risk, such as deep desaturations, must be balanced against a medium-term risk of hyperoxia and de-nitrogenation.

DETAILED DESCRIPTION:
Clearing the airways is a complex phenomenon involving the production of secretions, the nature of mucus (viscosity, elasticity, stringiness, and adhesiveness), ciliary movement, and coughing. Endotracheal suctioning are performed when the patient is "unable to clear the airways of obstructions hindering the free passage of air." Classically, endotracheal suctioning cause transient desaturation exacerbated by a decrease in cardiac output due to an increase in mean arterial pressure, promoting cardiac arrhythmias. To minimize these effects, it is recommended to perform additional preoxygenation, i.e., increasing the fraction of O2 in the air delivered to the patient by the ventilator 2-3 minutes before the procedure. These longstanding recommendations were reiterated in 2022, based on outdated studies involving systematic suctioning and/or disconnecting the patient from the ventilator.

Today, suctioning are performed on-demand, based on the patient's congestion status, either through the endotracheal tube cap or a "closed system." Desaturations have become rare without establishing that additional preoxygenation can prevent them. Moreover, additional preoxygenation is not without risks. In the short term, it induces de-nitrogenation atelectasis resulting in a loss of lung volume that can worsen pre-existing lung injuries in the most severe patients. In less severe cases, preoxygenation is responsible for transient hyperoxia, with various deleterious effects impacting patient prognosis. Thus, a short-term risk, such as deep desaturations, is juxtaposed with a medium-term risk of hyperoxia and de-nitrogenation.

The investigators hypothesize that the absence of additional preoxygenation is not inferior, in terms of deep desaturations, to the strategy with additional preoxygenation, and it would avoid exposing patients to the risks of de-nitrogenation-induced atelectasis and hyperoxia.

The investigators retained a margin of non-inferiority for the relative risk of 1.1, i.e. an increase of 10% of deep desaturations.

The main analysis will be performed on the per-protocol population (more conservative in non-inferiority trials).The per-protocol population will include patients who had at least one suctioning and for whom the additional preoxygenation strategy allocated by randomisation was followed in at least 70% of all suctioning reported in the patient's care record. Patients who stopped their participation in the study before endpoint timeframe and those who had never had an suctioning will not be included in the per protocol population.

The unit of analysis will be the patient, and a rate of suctioning leading to deep desaturation will be calculated for each patient, as described in the primary endpoint. The mean rate of suctioning leading to deep desaturation will then be calculated by treatment group (with additional preoxygenation / without additional preoxygenation).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Hospitalized in ICU, under invasive mechanical ventilation for less than 24 hours
* Information and signature of consent by patient or relative/trusted person, or emergency inclusion procedure

Exclusion Criteria:

* Patient on ECMO
* Not affiliated to a social security system
* Pregnant
* Under legal protection (curatorship, guardianship or safeguard of justice)
* Patient under AME
* Patient included in another interventional study that may have an impact on the evaluation criteria of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2260 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Rate of suctioning leading to deep desaturation | from Day 0 to ventilator weaning, and at the latest Day 28
  It will be calculated for each patient as the number of suctioning leading to deep desaturation (SpO2 88% or less, and 85% or less for patients with chronic obstructive pulmonary disease COPD), divided by the total number of endotracheal suctioning throughout the period. Oxygen saturation values will be collected every minute during the 15 minutes post-suctioning. Endotracheal suctioning in patients already ventilated with 100% FiO2 started prior to the decision to aspirate will not be taken into account

SECONDARY OUTCOMES:
Suctioning rate leading to severe desaturation | From Day 0 to ventilator weaning, and at the latest Day 28
  It will be calculated for each patient as the number of suctioning leading to severe desaturation (SpO2 85% or less, and 80% or less for patients with COPD), divided by the total number of endotracheal suctioning throughout the period
Number of ventilator free days at D28 | From Day 0 to Day 28
  Number of days without ventilation. In case of death value will be set to zero
Ventilator-associated pneumonia | From Day 0 to ICU-discharge, and at the latest Day 28
  Ventilator-associated pneumonia, as defined by the Formalized Recommendation of Experts from the SFAR-SRLF in 2017
Intensive care delirium | From Day 0 to ICU-discharge, and at the latest Day 28
  Delirium occurring in ICU, defined by a positive result on the CAM-ICU clinical assessment tool specific to ICU delirium
Composite criteria of ischemic phenomena in ICU, including one of the following: stroke, myocardial infarction, digestive ischemia | From Day 0 to ICU-discharge, and at the latest Day 28
  Composite criteria including at least one of the following: ischemic stroke, myocardial infarction, digestive ischemia
Ischemic stroke | From Day 0 to ICU-discharge, and at the latest Day 28
  Ischemic stroke occurring in intensive care, defined by the combination of the onset of focal motor deficit and compatible cerebral imaging
Myocardial infarction | From Day 0 to ICU-discharge, and at the latest Day 28
  Myocardial infarction occurring in intensive care, defined by an acute coronary syndrome with ST segment elevation and troponin elevation
Digestive ischemia | From Day 0 to ICU-discharge, and at the latest Day 28
  Digestive ischemia occurring in intensive care, diagnosed by CT scan or digestive endoscopy
Cardiac arrest | From Day 0 to ICU-discharge, and at the latest Day 28
  Cardiac arrest occuring in intensive care
Acute kidney injury | From Day 0 to ICU-discharge, and at the latest Day 28
  Acute kidney injury occurring in intensive care, defined by the initiation of renal replacement therapy
First bowel movements | From Day 0 to ICU-discharge, and at the latest Day 28
  Time to first bowel movements
ICU discharge vital status | At ICU discharge and at the latest Day 90
  Vital status at discharge from ICU
Hospital discharge vital status | At hospital discharge, and at the latest Day 90
  Vital status at discharge from hospital
Mean saturation over 15 minutes post-suctioning | From Day 0 to ventilator weaning, and at the latest Day 28
  Mean saturation over all the period of 15 minutes post suctioning
Absolute variation between saturation before suctioning and minimum saturation over 15 minutes post-suctioning | From Day 0 to ventilator weaning, and at the latest Day 28
  Saturation over all the period of 15 minutes post suctioning
Acute respiratory distress syndrome (ARDS) | From Day 0 to hospital discharge, and at the latest Day 90
  ARDS according to the Berlin definition, characterized by 1) acute respiratory failure evolving for a week or less, 2) bilateral opacities on thoracic imaging, 3) no evidence of predominant hydrostatic edema, 4) hypoxemia with a PaO2/FIO2 ratio < 300 mmHg for positive end-expiratory pressure set at 5 cmH2O or more, with 3 severity stages defined based on hypoxemia
Length of ICU stay | at ICU discharge, and at the latest Day 90
  Length of stay in intensive care
Length of hospital stay | at hospital discharge, and at the latest Day 90
  Length of stay in hospital
Time in minutes between endotracheal suctioning and eventual desaturation | From Day 0 to ventilator weaning, and at the latest Day 28
  For each desaturation, time in minutes between endotracheal suctioning and desaturation

CONTACTS AND LOCATIONS:
Overall Officials: Claire FAZILLEAU, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.